CLINICAL TRIAL: NCT01013376
Title: A Pilot, Single-Center, Open-Label Study of the Safety of MC-1101 in Both Normal Volunteers and Patients With Early Non-exudative Age-Related Macular Degeneration
Brief Title: A Pilot Study of the Safety of MC-1101 in Both Normal Volunteers and Patients With Early Dry AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacuCLEAR, Inc. (Industry)
Responsible Party: Philip G. Ralston, Jr. / President & CEO, MacuCLEAR, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1101-CBF-01
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Topical administration of MC-1101
  Interventions: Drug: MC-1101
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: MC-1101 — MC-1101 1.0%
  Arms: Active
Drug: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
The safety and comfort of repeated administrations of a topically-administered ophthalmic formulation of MC-1101 will be established through investigator assessments and subject reporting over a 3 day period. Safety assessments will be performed on both normal, healthy subjects as well as those with the signs and symptoms of early non-exudative age-related macular degeneration (dry AMD).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of dry AMD or;
* Normal, healthy volunteer

Exclusion Criteria:

* Uncontrolled systemic disease
* Women who are pregnant, nursing, or planning a pregnancy during the study's duration

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Ocular safety | 3 days

SECONDARY OUTCOMES:
Choroidal blood flow assessment | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Torkildsen, M.D., Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States